CLINICAL TRIAL: NCT04003168
Title: A Phase I Clinical Trial to Evaluate the Safety and Efficacy of Human BCMA Targeted T Cells Injection for Subjects With BCMA-positive Relapsed/Refractory Multiple Myeloma
Brief Title: Human BCMA Targeted T Cells Injection Therapy for BCMA-positive Relapsed/Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai Changzheng Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN01-MM01
Record Dates: First submitted 2019-06-24; First posted 2019-07-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Multiple Myeloma
Keywords: BCMA; CAR-T; multiple myeloma; Relapsed/Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human BCMA targeted T Cells Injection (Experimental): A single infusion of anti-BCMA CAR transduced T cells administered intravenously at a target dose of 3 to 9 x 10^6 CAR T +cells/kg. The classic "3+3" dose escalation will be applied.
  Interventions: Drug: Human BCMA targeted T Cells Injection

INTERVENTIONS:
Drug: Human BCMA targeted T Cells Injection — Autologous genetically modified anti-BCMA CAR transduced T cells

SUMMARY:
To evaluate the safety and efficacy of Human BCMA Targeted T Cells Injection for the treatment of BCMA-positive relapsed/refractory multiple myeloma. Patients will be given a conditioning chemotherapy regimen of fludarabine and cyclophosphamide followed by a single infusion of BCMA CAR+ T cells.

DETAILED DESCRIPTION:
Participants with BCMA-positive relapsed/refractory multiple myeloma can participate if all eligibility criteria are met. Tests required to determine eligibility include disease assessments, a physical exam, Electrocardiograph, CT/MRI/PET, and blood draws. Participants receive chemotherapy prior to the infusion of BCMA CAR+ T cells. After the infusion, participants will be followed for side effects and effect of BCMA CAR+ T cells. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects volunteer to participate in clinical research, understand and know the research and sign informed consent document, willing to complete all the trial procedures;
2. 18 to 70 Years Old, Male and female;
3. Expected survival > 12 weeks;
4. Previously diagnosed as multiple myeloma by IMWG updated criteria (2014);
5. Patients with positive pathological test results or flow cytometry proving that BCMA expression of malignant plasma cells in bone marrow or plasma cell tumors ≥30%;
6. One of the following indicators is satisfied:

   1. Serum M protein IgG ≥ 10 g/L, or IgA > 10 mg/L, or IgD > 5 mg/L;
   2. Urine M protein ≥ 200 mg/24h;
   3. Serum free light chain ≥ 100 mg/L;
7. Patients with relapsed/refractory multiple myeloma. Relapsed is defined as:

   Patients have disease progression after at least three-line treatment regimens. Patients previously received at least 3 different mechanisms treatment regimens for multiple myeloma, including protease inhibitors and immunomodulators, and have disease progression within 60 days of the latest treatment ; Refractory is defined as: Patients who achieved remission in the piror therapies, have disease progression within 60 days, or after the latest therapy.
8. Those who relapse 90 days after stem cell transplantation
9. ECOG score 0-1;
10. Liver, kidney and cardiopulmonary functions meet the following requirements:

    1. Creatinine clearance (estimated by Cockcroft Gault formula) ≥ 40 mL/min;
    2. Left ventricular ejection fraction >50%;
    3. Baseline peripheral oxygen saturation >95%;
    4. Total bilirubin ≤ 2×ULN; ALT and AST ≤2.5 × ULN;
11. The venous access required for collection can be established, and no leukocyte collection contraindications.

Exclusion Criteria:

1. Accompanied by other uncontrolled malignancies;
2. Subjects with positive HBsAg or HBcAb and peripheral blood HBV DNA titer is higher than the lower limit of detection of the research institution; HCV antibody positive and peripheral blood HCV RNA positive; HIV antibody positive; syphilis primary screening antibody positive;
3. Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), severe arrhythmia, liver, kidney or metabolic disease with poor drug control;
4. Patients who are accounted to be not appropriate for this trail by investigator;
5. Pregnant or lactating, or planning to have a pregnancy during or within 1 year after treatment;
6. Received CAR-T treatment or other gene therapies before enrollment;
7. Those who failed to sign informed consent form or comply with the research procedures; Unwilling or unable to comply with research requirements;
8. Have had severe immediate hypersensitivity reactions to any drugs used in this research;
9. The presence or suspicion of fungi, bacteria, viruses or other infections that are uncontrollable or requiring intravenous treatment;
10. In the past two years, the terminal organ was damaged due to autoimmune diseases (such as crohn's disease, rheumatoid arthritis, systemic lupus erythematosus), or the systemic use of immunosuppressive or other systemic disease control drugs was required;
11. Have a history of central nervous system (CNS) disease, such as epilepsy, seizures, paralysis, aphasia, stroke, severe brain damage, dementia, Parkinson's disease, psychosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE 5.0 | 28 days post infusion

SECONDARY OUTCOMES:
Concentration of Anti-BCMA CAR T Cells in blood | 2 years post infusion
Concentration of Anti-BCMA CAR T Cells in bone marrow | 2 years post infusion
Pharmacodynamics (Levels of Cytokines in Serum) | 2 years post infusion
Pharmacodynamics (Content of clonal plasma cells in bone marrow) | 2 years post infusion
Overall response rate (ORR) after administration | 3 months post infusion
Negative proportion of minimal residual disease (MRD) | 28 days post infusion
Duration of remission (DOR) after administration | 2 years post infusion
Progress Free Survival (PFS) after administration | 2 years post infusion
Overall Survival (OS)after administration | 2 years post infusion
Positive incidence of anti-drug antibody | 2 years post infusion

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Wang H, Tsao ST, Gu M, Fu C, He F, Li X, Zhang M, Li N, Hu HM. A simple and effective method to purify and activate T cells for successful generation of chimeric antigen receptor T (CAR-T) cells from patients with high monocyte count. J Transl Med. 2022 Dec 19;20(1):608. doi: 10.1186/s12967-022-03833-6. PMID 36536403